CLINICAL TRIAL: NCT04150120
Title: eHealth as an Aid for Facilitating and Supporting Self-management in Families With Long-term Childhood Illness - Development, Evaluation and Implementation in Clinical Practice
Brief Title: eHealth as an Aid for Facilitating and Supporting Self-management in Families With Long-term Childhood Illness
Acronym: eChildHealth
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Lund University (Other)
Collaborators: Skane University Hospital (Other); Rigshospitalet, Denmark (Other); Arba Minch University (Other); University of Iceland (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2018-01399
Record Dates: First submitted 2019-10-21; First posted 2019-11-04 (Actual); Last update posted 2022-12-09 (Actual); Status verified 2022-12

CONDITIONS: Preterm Birth; Pediatric Cancer; Hirschsprung Disease; Congenital Malformation; Congenital Heart Disease; Nutrition Disorder, Child
Keywords: e-health; children; culture; health economy; quality of life; home care
MeSH Terms: conditions — Premature Birth; Neoplasms; Hirschsprung Disease; Congenital Abnormalities; Heart Defects, Congenital; Child Nutrition Disorders

STUDY DESIGN:
Intervention Model Description: Consecutive series of legal guardians to children fulfilling the inclusion criteria in each arm. The legal guardians will be asked to 1) be involved in the development of the eHealth application, 2) evaluate the eHealth application at home, or 3) serve as a control group receiving traditional follow-up after discharge.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Reconstructive paediatric surgery (Area I) (Active Comparator): The overall incidence of congenital malformations in the gastrointestinal and urinary tract needing surgical interventions is about 1:1000 (Swedish national malformation registers) with a morbidity during childhood about 20-60%. Advanced paediatric surgery for the diagnosis Hirschsprung's disease, anorectal malformations, bladder extrophy, congenital diaphragmal hernia, and esophageal atresia is from July 2018 only performed at two NCSM in Sweden. The NCSM at Skåne University Hospital (SUS) in Lund forms one context. The quality of postoperative care is of immense importance both for short and long-term outcome. Legal guardians describe their situation after leaving the hospital as extremely stressful as they have not only to take responsibility for their new-born child but also of surgical wounds, medications, treatments, and special nutritional needs.
  Interventions: Device: e-health device with application
- Congenital heart disease (Area II) (Active Comparator): In Sweden, about 8-10 in 1000 children per year are born with congenital heart disease (CHD). CHD is a birth defect that leads to frequent hospitalisation, long hospital stays, and extreme anxiety for parents (18). In Sweden, paediatric heart surgery is concentrated to two NCSM of which one is situated at SUS, Lund where 250-300 children have cardiac surgery every year. Children with complicated CHD require contact and follow-up visits for a long time after the heart surgery and many families have to travel long for surgery (for example from Iceland), postoperative care and follow-up visits. Telemedicine after reconstructive cardiac surgery in children is shown to be feasible, although challenging and reduced unscheduled visits.
  Interventions: Device: e-health device with application
- Preterm born (Area III) (Active Comparator): Most prematurely born children grow up to be healthy, but as a group, they are at a greater risk of developing cognitive, emotional and behavioural problems. Every year 7% of all children are born prematurely (gestational age of less than 37 weeks) and the numbers of preterm births are rising in Sweden as well as internationally. Preterm births often involve long hospitalisations for children and parents, and discharge from the hospital often means a difficult transition for parents in both short and long-term perspectives. Traditionally, communication with parents following discharge has been through home visits or telephone calls. By communicating through digital technology, it may be possible to improve the support to parents and thereby make the transition from hospital to home less stressful.
  Interventions: Device: e-health device with application
- Paediatric oncology (Area IV) (Active Comparator): For children with cancer, treatment and follow-up at home is common. At the same time, families wish to minimize the negative impact on family members' social and everyday life. Home medication management is a high-risk area and medication errors are common, particularly among parents of children with cancer. Thus, parents are responsible for complex care and regular follow-up in their home with an increased need for education as well as clinical management support. At present, there are no, or limited, professional outreach support to support them and their families. Communication with parents following discharge has been through e-mail and/ or telephone calls. By communicating through digital technology, it may be possible to improve the support to children and parents.
  Interventions: Device: e-health device with application
- Intravenous infusion therapy at home (Area V) (Active Comparator): For children with LTI administration of intravenous infusion therapy at home is an increasingly important area. Home medication management is a high-risk area and medication errors are common, particularly among parents of children with cancer. Thus, parents are responsible for complex care in their home with an increased need for educational as well as clinical management support during home infusion therapy. At present, children and adolescents with LTI at the University Hospital of Copenhagen receive home infusion therapy by a portable pump with no assistance from an outreaching team to support them and their families.
  Interventions: Device: e-health device with application
- Children with cerebral palsy (VI) (Active Comparator): Cerebral palsy (CP) is the most common physical disability in childhood. Approximately 2-2.5/1000 children have CP with affected muscle tone, movement and motor skills, often accompanied by pain, epilepsy and intellectual, communicational and behavioural impairment. Early detection is challenging but important for minimizing the consequences from neurodevelopmental impairment by an early and right treatment. General Movement Assessment (GMA), an observational method for classification of spontaneous movements in young infants, is currently the most accurate method for early identification of CP. Video recordings are taken with a standardised video set-up in the hospitals regular follow-up clinics when the child is 10 to 20 weeks post-term age. Performing video recordings at home by the parents at a time, which suits the family and the child, would optimize the chances for a successful recording.
  Interventions: Device: e-health device with application

INTERVENTIONS:
Device: e-health device with application — In this project we focus on eHealth solutions for patients and/or their families in situations where they could benefit from enhanced communication options with specialist staff. In this design space we use a model where a 4G-enabled tablet computer is lent to the families for the length of the study, thus avoiding economic requirements on the families and keeping the equipment uniform. The tablets run an application that enables multiple forms of direct and bi-directional communication in real-time with specialist staff at the hospital. For the staff, the technical situation is different; here we have in earlier demonstrators used web-based solutions accessed with existing computer equipment.

SUMMARY:
The overall aim is twofold: 1) to stretch the borderline regarding the present knowledge of clinical and economic cost-effectiveness of eHealth as an aid for facilitating and supporting self-management in families with long-term childhood illness, and 2) to develop a sustainable multidisciplinary research environment for advancing, evaluating, and implementing models of eHealth to promote self-management for children and their families.

A number of clinical studies are planned for, covering different parts of paediatric healthcare. The concept of child-centred care is essential. Experienced researchers from care science, medicine, economics, technology, and social science will collaborate around common issues. Expertise on IT technology will analyse the preconditions for using IT; economic evaluations will be performed alongside clinical studies; and cultural and implementation perspectives will be used to analyse the challenges that arise from the changes in relations among children, family and professionals, which may occur as a result of the introduction of eHealth.

Child health is not only important in itself. Investments in child health may also generate significant future gains, such as improved educational and labour market performance. Six complex, long-term and costly challenges in paediatric healthcare are planned for, involving eHealth technology such as interactive video consultation, pictures, on-line monitoring, and textual communication. The research follows an international framework for developing and evaluating complex interventions in healthcare. End-users (families) and relevant care providers (professionals in health and social care) will participate throughout the research process. The overall aim is certainly to analyse eHealth as an aid for facilitating and supporting self-management. However, the plan also includes the research issue whether eHealth at the same time improves the allocation of scarce health care- and societal resources.

DETAILED DESCRIPTION:
The vision for the coming 6-year period is to establish multi-disciplinary research, designed to strengthen and advance the knowledgebase of eHealth as an aid for facilitating and supporting self-management among children with long-term illness and their families. The programme builds on interventions and implementation in three research domains: (1) eHealth to enable and promote self-management in advanced paediatric care, (2) eHealth for early diagnosis and treatment in paediatric healthcare, and (3) Co-creation of multi-disciplinary knowledge for the translation of eHealth in practice.

The overall goals of the research programme are to:

Evaluate, advance and implement models of eHealth to improve self-management for children and adolescents with or at risk for long-term illness and their families for better allocation of family-, healthcare- and societal resources.

Increase the knowledge of cultural factors and implementation strategies to facilitate implementation processes in general, and more specifically generate theoretical and methodological models on how to successfully implement eHealth in paediatric care.

Enhance the translation and integration of new research findings within eHealth into care services and the wider society by supporting healthcare professionals in their provision of evidence-based care and by translating and communicating research results to them as well as stakeholders and families.

Enhance the research proficiency of junior researchers in paediatric care and eHealth nationally and internationally through collaborative approaches in both inter- and multidisciplinary groups.

Two features of healthcare systems today are easily detected: 1) a trend towards more reliance on the individual and family to take active part in the healthcare process - with self-management being a keyword, and 2) great expectations regarding the potential benefits of using modern information technology in the domain of health and health care. The complex and costly needs for care of an increasing number of children with long-term illness (LTI) i.e. an illness that lasts for three months or more, generally has a slow progression, and can be controlled but not cured [1]) is one of the most critical challenge for healthcare systems all over the world. In addition to poorer health, people with LTI generally have lower educational achievements, fewer economic opportunities, and higher rates of poverty. Ensuring healthy growth and development in children is a principal concern of all societies. In this context, eHealth is of special interest as an aid for facilitating and supporting self-management for children with and at risk for LTI.

Self-management is the use of own time and money for individual and family health promotion. It is an ingredient in almost all measures for promoting health. Pure self-management in health relies on own efforts without formal intervention of health care services. On the other extreme, there are formal healthcare activities that require 100 percent of healthcare inputs for example surgery under anaesthesia. In most instances, both types of inputs are necessary - in varying degrees. The choice of self-management activities and its results depend on family-member preferences, knowledge, and attitudes. In order for healthcare system initiatives to be accepted and successful, they must be attuned to these characteristics. Individual tailoring is all the more important, the more reliance is on self-management. Thus, in the process of developing and evaluating new treatment modes, user participation is essential.

eHealth is a broad concept as indicated by the WHO definition: "eHealth is the transfer of health resources and healthcare by electronic means", i.e. also including older techniques such as telemedicine. Great expectations are associated with the realisation of the term. It may: 1) increase communication between healthcare providers and patients, 2) increase accessibility and patient participation in healthcare, and 3) support information and data sharing between patients, family and health-service providers http://www.euro.who.int/en/ehealth. It might be observed that the term eHealth does not preclude the use of electronic means to improve communication between providers within the healthcare system, potentially increasing the internal efficiency of formal healthcare, without any direct effects on patients and families. Here, however, the focus is on the role of eHealth as an aid for facilitating and supporting self-management, i.e. a concern with a wider, societal perspective on the allocation of scarce resources for health.

Cost-effectiveness is one of the ethical principles that are supposed to govern decisions on the allocation of scarce healthcare resources in Sweden. Thus, new healthcare technology should not be introduced if not proven cost-effective in comparison to existing (best) practice. Requirements for the economic evaluation of new healthcare technology exist in most Western countries. To date, economic evaluations of eHealth reported in the literature are scare and suffer from lack of randomised control trials (RTCs), small sample sizes, and the absence of high-quality data or appropriate measures.

Paediatric healthcare is rapidly evolving towards outpatient and community-care and from public to parental responsibility. This form of care is however rarely backed-up with communication support. In Sweden and most Western countries, highly specialised paediatric healthcare is confined to few National Centres of Specialized Medicine (NCSM) http://www.socialstyrelsen.se/rikssjukvard. This means that following birth a large majority of children with congenital malformations are transported to hospitals far away from home for advanced surgery. Following discharge, the outermost medical and nursing competence for the child will be at the NCSM. International policy and practice aim for infants, older children and adolescents with LTI to be cared for at home as much as possible to reduce the distress of hospital admissions and to keep up the normal family life. Limited research exists on the effect of digital interactive care on parents and children. eHealth in the home setting is often preferred by parents, especially by parents of newborns but has still not been widely adopted. Digital techniques can aid safer post-operative healthcare at home and may reduce costs to patients and society. This in turn might lead to more confident use of self-management and an increased sense of security at home. In some areas in paediatric care telemedicine initiatives is shown to benefit resources, enrich the community, and improve care that ultimately serve to better patient health.

Six clinical research projects are planned, illustrating complex, highly specialized, often long-term and costly decision-making challenges in paediatric care, for developing, evaluating implementing, and utilising different devices of eHealth technology. In addition, four more research projects will be performed in parallel to provide general analyses of eHealth in paediatric care and to facilitate and support economic, technical, cultural, and organisational analyses of the clinical data.

Bridging the hospital care and safe care at home for children with LTI with the aid of eHealth is a vital clinical area, especially for professionals in nursing, physiotherapy and medicine. However, also for the scientific area in health science it is of great importance as eHealth change the communication between children, parents and health professionals. This is a new research area that needs to be explored.

To develop, evaluate and implement eHealth devices in clinical care, an inter- and multidisciplinary approach is needed. Therefore, the investigators well-functioning and long-lasting clinical and research collaboration in health science, medicine, global health, health economics, technology, and social science has been enhanced to respond to the needs in paediatric care. Thereby, it is possible to address the important study of encounters with technology and various methods of communications and how eHealth aid can capture complex exchange of wellbeing and health, and feelings and perceptions of for example anxiety, stress levels, safety, many of which are culturally related. Also, values and contexts are sensitive to communication methods. The studies will therefore contribute significantly to the research area of eHealth as an aid for facilitating and supporting self-management in paediatric care, but not only. The programme also includes the research issue whether eHealth at the same time improves the allocation of scarce healthcare- and societal resources.

The multi-method design including both qualitative and quantitative methods will enhance the understanding to advance and evaluate routines and practices for better physiological and psychological outcomes in children with LTI and their families. The clinical projects will also contribute to a deeper understanding on identifying risk factors for complications and how to prevent adverse events in care performed at home.

In this programme, the focus is on eHealth solutions for situations where children and their families can be supported by enhanced communication for self-management with specialist professionals most commonly with specialist nurses. In such situations, it is important to find technical solutions that are both easy to use for all involved, easily accessible for families, and efficient to use for the professionals. Design options include web browser-based solutions, application-based solutions for larger mobile devices such as touchpads and application for mobile phones while observing the strict security rules for personal health information. An issue of accessibility is also to avoid economic demands on e.g. families not having access to appropriate equipment. Furthermore, relying on patient's equipment increases the technical demand and testing as the variation of equipment is huge, while the number of patients is comparatively small. Typically, technologies and applications develop at a high pace driven by commercial interests and may not be synchronised with a corresponding development of the understanding of possibilities and limitations of the applications in specific areas of care.

Importantly, the studies within different clinical contexts and considering cost-effectiveness, technical development, cultural and implementation aspects contribute to the knowledge and understanding about how eHealth can reduce the information asymmetry between providers, developers and consumers for further implementation into clinical practices, policies, and procedures. This programme also provides a significant contribution to a grounded and evidence-based understanding of both possibilities and limitations of eHealth applications in this area not only in terms of their efficacy but also in terms of the possible ethical conflicts involved in the introduction of new technology.

ELIGIBILITY:
Inclusion Criteria (Intervention group):

Legal guardians of children below four years of age who are hospitalised for:

* reconstructive surgery for congenital malformations
* cardiac surgery for CHD
* premature birth
* paediatric cancer and in treatment
* are in need of nutritional supplements
* are about to be discharged from the hospital
* are able to communicate in the local language (Swedish in Sweden and Danish in Denmark)
* signs informed consent

Inclusion Criteria (Control group):

Legal guardians of children below four years of age who fulfil the intervention group inclusion criteria but:

* do not want to use the e-device
* not recruited for the intervention group
* are recruited after the stipulated numbers for the intervention group are met

Exclusion Criteria:

* Legal guardians of children fulfilling the inclusion criteria but where the child has complications or comorbidity which may affect the results of the study (as defined by the responsible medical physician)
* The legal guardian refuses to sign informed consent.

Ages: 3 Days to 47 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 420 (Estimated)
Dates: Start 2019-10-15 (Actual); Primary Completion 2024-10-15 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
The PedsQL Healthcare Satisfaction Generic Module | After their participation in the study has ended, on average after 2-4 weeks.
  The PedsQL Healthcare Satisfaction Generic Module is composed of 24 items comprising 6 dimensions. Item scaling: 5-point Likert scale: 0 (Never) to 4 (Always) and Not Applicable. Higher scores indicate higher satisfaction. The scale includes the variables: information, family inclusion, communication, technical skills, emotional needs, and overall satisfaction.
Cost-utility ratios | After their participation in the study has ended, on average after 2-4 weeks.
  Health economic variables

SECONDARY OUTCOMES:
The child's general and specific health status | Before the study begins and after their participation in the study has ended, on average after 2-4 weeks.
  This questionnaire contains information about the health of each child both at the time when the study begins and when the study ends. It asks for information on the weight of the child, the diagnosis, the treatment, specific needs when released from hospital, general health status when released from hospital, general health status at end of study. The answers are either given as multiple choice or as free text.
The PedsQL 2.0 Family Impact Module | After their participation in the study has ended, on average after 2-4 weeks.
  The PedsQL 2.0 Family Impact Module is composed of 36 items comprising 8 dimensions. Item scaling: 5-point Likert scale: 5-point Likert scale from 0 (Never) to 4 (Almost always). Higher scores indicate better functioning.
The Parental Stress (Parental - Persistent Role Problems) | After their participation in the study has ended, on average after 2-4 weeks.
  The Parental Stress (Parental - Persistent Role Problems) is composed of 9 items. Item scaling: 5-point Likert scale: 5-point Likert scale from 0 (Does not happen) to 4 (Happens always). Lower scores indicate less stress.
Adverse events that occurs during the study period | After their participation in the study has ended, on average after 2-4 weeks.
  Any adverse events occurring during the study period will be recorded in free text format by the staff for all participants.
The Clavien-Dindo Classification | After their participation in the study has ended, on average after 2-4 weeks.
  The therapy used to correct a specific complication is the basis of this classification in order to rank a complication in an objective and reproducible manner. The scale consists of 7 grades (I, II, IIIa, IIIb, IVa, IVb and V). A high grade indicates a more severe problem.
Length of hospital stay | After their participation in the study has ended, on average after 2-4 weeks.
  Days
Number of routine and acute visits | After their participation in the study has ended, on average after 2-4 weeks.
  Number of routine and acute visits
Health economic variables: Family time | After their participation in the study has ended, on average after 2-4 weeks.
  Distribution of family time use
Health economic variables: Family economy | After their participation in the study has ended, on average after 2-4 weeks.
  Family economy
Health economic variables: Hopsital resources | After their participation in the study has ended, on average after 2-4 weeks.
  Use of hospital resources
Health economic variables: Health care resources | After their participation in the study has ended, on average after 2-4 weeks.
  Use of other healthcare resources
Health economic variables: Health care expenditures | After their participation in the study has ended, on average after 2-4 weeks.
  Healthcare expenditures by type of resource
Health economic variables: Productivity | After their participation in the study has ended, on average after 2-4 weeks.
  Loss of production
Health economic variables: Utility | After their participation in the study has ended, on average after 2-4 weeks.
  Utility scores.
EQ-5D-3L | After their participation in the study has ended, on average after 2-4 weeks.
  The EQ-5D-3L descriptive system comprises the following five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 levels: no problems, some problems, and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results into a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.

CONTACTS AND LOCATIONS:
Overall Officials: Inger Kristensson Hallström, PhD, Principal Investigator — Lund University
Locations (6):
- Denmark (2):
  - Rigshospitalet, Copenhagen
  - Hillerød Hospital, Hillerød
- Sweden (4):
  - Neonatal Department, Skåne University Hospital, Lund, Skåne County
  - Paediatric Cardiology Department, Skåne University Hospital, Lund, Skåne County
  - Paediatric Oncology Department, Skåne University Hospital, Lund, Skåne County
  - Paediatric Surgery Department, Skåne University Hospital, Lund, Skåne County

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Perrin EC, Newacheck P, Pless IB, Drotar D, Gortmaker SL, Leventhal J, Perrin JM, Stein RE, Walker DK, Weitzman M. Issues involved in the definition and classification of chronic health conditions. Pediatrics. 1993 Apr;91(4):787-93. PMID 8464668
- [Background] World report on disability. 2011; Available from: http://www.who.int/disabilities/world_report/2011/en/.
- [Background] Grossman, M., The Determinants of Health: An Economic Perspective. 2017, New York: Columbia University Press
- [Background] Chan CV, Kaufman DR. A framework for characterizing eHealth literacy demands and barriers. J Med Internet Res. 2011 Nov 17;13(4):e94. doi: 10.2196/jmir.1750. PMID 22094891
- [Background] de la Torre-Diez I, Lopez-Coronado M, Vaca C, Aguado JS, de Castro C. Cost-utility and cost-effectiveness studies of telemedicine, electronic, and mobile health systems in the literature: a systematic review. Telemed J E Health. 2015 Feb;21(2):81-5. doi: 10.1089/tmj.2014.0053. Epub 2014 Dec 4. PMID 25474190
- [Background] Parab CS, Cooper C, Woolfenden S, Piper SM. Specialist home-based nursing services for children with acute and chronic illnesses. Cochrane Database Syst Rev. 2013 Jun 15;2013(6):CD004383. doi: 10.1002/14651858.CD004383.pub3. PMID 23771694
- [Background] Tan K, Lai NM. Telemedicine for the support of parents of high-risk newborn infants. Cochrane Database Syst Rev. 2012 Jun 13;2012(6):CD006818. doi: 10.1002/14651858.CD006818.pub2. PMID 22696360
- [Background] Danbjorg DB, Wagner L, Kristensen BR, Clemensen J. Intervention among new parents followed up by an interview study exploring their experiences of telemedicine after early postnatal discharge. Midwifery. 2015 Jun;31(6):574-81. doi: 10.1016/j.midw.2015.02.007. Epub 2015 Feb 24. PMID 25765743
- [Background] Bradford NK, Young J, Armfield NR, Herbert A, Smith AC. Home telehealth and paediatric palliative care: clinician perceptions of what is stopping us? BMC Palliat Care. 2014 Jun 16;13:29. doi: 10.1186/1472-684X-13-29. eCollection 2014. PMID 24963287
- [Background] Marklund B, Strom M, Mansson J, Borgquist L, Baigi A, Fridlund B. Computer-supported telephone nurse triage: an evaluation of medical quality and costs. J Nurs Manag. 2007 Mar;15(2):180-7. doi: 10.1111/j.1365-2834.2007.00659.x. PMID 17352701
- [Background] Stone JM, Gibbons TE. Telemedicine in Pediatric Gastroenterology: An Overview of Utility. Telemed J E Health. 2018 Aug;24(8):577-581. doi: 10.1089/tmj.2017.0234. Epub 2017 Dec 22. PMID 29271722
- [Background] Mansson C, Jakobsson U, Lundqvist P. Translation and psychometric evaluation of a Swedish version of the parental stressor scale PSS: NICU. Scand J Caring Sci. 2016 Mar;30(1):193-201. doi: 10.1111/scs.12217. Epub 2015 Apr 28. PMID 25918977
- [Background] Hansson H, Kjaergaard H, Johansen C, Hallstrom I, Christensen J, Madsen M, Schmiegelow K. Hospital-based home care for children with cancer: feasibility and psychosocial impact on children and their families. Pediatr Blood Cancer. 2013 May;60(5):865-72. doi: 10.1002/pbc.24474. Epub 2013 Jan 17. PMID 23335455
- [Background] Tiberg, I., The initial care when a child is diagnosed with type 1 diabetes. Doctoral dissertation series /Faculty of Medicine, Lund University: 2012:48. 2012: Lund : Faculty of Medicin, Lund University, 2012.
- [Background] Graneli C, Dahlin E, Borjesson A, Arnbjornsson E, Stenstrom P. Diagnosis, Symptoms, and Outcomes of Hirschsprung's Disease from the Perspective of Gender. Surg Res Pract. 2017;2017:9274940. doi: 10.1155/2017/9274940. Epub 2017 Mar 7. PMID 28367493
- [Background] Ost E, Nisell M, Frenckner B, Mesas Burgos C, Ojmyr-Joelsson M. Parenting stress among parents of children with congenital diaphragmatic hernia. Pediatr Surg Int. 2017 Jul;33(7):761-769. doi: 10.1007/s00383-017-4093-4. Epub 2017 May 19. PMID 28527042
- [Background] Miller GG, Levesque K. Telehealth provides effective pediatric surgery care to remote locations. J Pediatr Surg. 2002 May;37(5):752-4. doi: 10.1053/jpsu.2002.32270. PMID 11987093
- [Background] Hearps SJ, McCarthy MC, Muscara F, Hearps SJ, Burke K, Jones B, Anderson VA. Psychosocial risk in families of infants undergoing surgery for a serious congenital heart disease. Cardiol Young. 2014 Aug;24(4):632-9. doi: 10.1017/S1047951113000760. Epub 2013 Jun 27. PMID 23803336
- [Background] Black AK, Sadanala UK, Mascio CE, Hornung CA, Keller BB. Challenges in implementing a pediatric cardiovascular home telehealth project. Telemed J E Health. 2014 Sep;20(9):858-67. doi: 10.1089/tmj.2013.0343. Epub 2014 Aug 1. PMID 25083905
- [Background] Lundqvist, P., Children born prematurely : their fathers' experiences and trends in mortality and morbidity during a ten-year period. Lund University, Faculty of Medicine doctoral dissertation series: 2008:117. 2008: Lund : Lund University, 2008.
- [Background] Hall, E.C.O., et al., The journey towards motherhood after a very preterm birth: Mothers' experiences in hospital and after home-coming. Journal of Neonatal Nursing, 2013. 19(3): p. 109-113.
- [Background] Walsh KE, Roblin DW, Weingart SN, Houlahan KE, Degar B, Billett A, Keuker C, Biggins C, Li J, Wasilewski K, Mazor KM. Medication errors in the home: a multisite study of children with cancer. Pediatrics. 2013 May;131(5):e1405-14. doi: 10.1542/peds.2012-2434. Epub 2013 Apr 29. PMID 23629608
- [Background] Novak I, Hines M, Goldsmith S, Barclay R. Clinical prognostic messages from a systematic review on cerebral palsy. Pediatrics. 2012 Nov;130(5):e1285-312. doi: 10.1542/peds.2012-0924. Epub 2012 Oct 8. PMID 23045562
- [Background] Brown AK, Greisen G, Haugsted U, Jonsbo F. Formal training in general movement assessment is required to effectively evaluate infants with perinatal asphyxia in outpatient settings. Acta Paediatr. 2016 Sep;105(9):1056-60. doi: 10.1111/apa.13491. Epub 2016 Jun 24. PMID 27240948
- [Background] Biru M, Hallstrom I, Lundqvist P, Jerene D. Rates and predictors of attrition among children on antiretroviral therapy in Ethiopia: A prospective cohort study. PLoS One. 2018 Feb 6;13(2):e0189777. doi: 10.1371/journal.pone.0189777. eCollection 2018. PMID 29408897
- [Background] Bolin K, Jacobson L, Lindgren B. The family as the health producer--when spouses are Nash-bargainers. J Health Econ. 2001 May;20(3):349-62. doi: 10.1016/s0167-6296(00)00086-2. PMID 11373835
- [Background] Kristjansdottir O, Unruh AM, McAlpine L, McGrath PJ. A systematic review of cross-cultural comparison studies of child, parent, and health professional outcomes associated with pediatric medical procedures. J Pain. 2012 Mar;13(3):207-19. doi: 10.1016/j.jpain.2011.12.008. PMID 22386060
- [Background] Flores G; Committee On Pediatric Research. Technical report--racial and ethnic disparities in the health and health care of children. Pediatrics. 2010 Apr;125(4):e979-e1020. doi: 10.1542/peds.2010-0188. Epub 2010 Mar 29. PMID 20351000
- [Background] Ross J, Stevenson F, Lau R, Murray E. Factors that influence the implementation of e-health: a systematic review of systematic reviews (an update). Implement Sci. 2016 Oct 26;11(1):146. doi: 10.1186/s13012-016-0510-7. PMID 27782832
- [Background] Craft MJ, Willadsen JA. Interventions related to family. Nurs Clin North Am. 1992 Jun;27(2):517-40. PMID 1584702
- [Background] Craig P, Dieppe P, Macintyre S, Michie S, Nazareth I, Petticrew M; Medical Research Council Guidance. Developing and evaluating complex interventions: the new Medical Research Council guidance. BMJ. 2008 Sep 29;337:a1655. doi: 10.1136/bmj.a1655. PMID 18824488
- [Background] Johannesson. and Perjsons., An Introduction to Design Science. 2014: Springer.
- [Background] Creswell, J. and V. Plano Clark, Designing and conducting mixed methods research. 2011, Thousand Oaks, CA: Sage.
- [Background] Coyne I, Hallstrom I, Soderback M. Reframing the focus from a family-centred to a child-centred care approach for children's healthcare. J Child Health Care. 2016 Dec;20(4):494-502. doi: 10.1177/1367493516642744. Epub 2016 Jul 25. PMID 27141084
- [Background] Weiss, D. and C. Marmar, Assessing Psychological Trauma and PTSD in The Impact of Event Scale-Revised, W. JP and K. TM, Editors. 1997, Guilford Press: New York. p. 399-411.
- [Background] Abidin, R., Parenting Stress Index, in Professional Manual. 1995, Psychological Assessment Resources, Inc: Odessa.
- [Background] Norman CD, Skinner HA. eHEALS: The eHealth Literacy Scale. J Med Internet Res. 2006 Nov 14;8(4):e27. doi: 10.2196/jmir.8.4.e27. PMID 17213046
- [Background] Damschroder LJ, Lowery JC. Evaluation of a large-scale weight management program using the consolidated framework for implementation research (CFIR). Implement Sci. 2013 May 10;8:51. doi: 10.1186/1748-5908-8-51. PMID 23663819
- [Background] Berry, J.W., et al., Cross-cultural psychology: Research and applications. 3 ed. 2011, Cambridge, UK: Cambridge Univ Press.
- [Background] Chernick, M., Bootstrap Methods: A Practitioner's Guide. . 1999, New York: John Wiley & Sons.
- [Background] Graneheim UH, Lundman B. Qualitative content analysis in nursing research: concepts, procedures and measures to achieve trustworthiness. Nurse Educ Today. 2004 Feb;24(2):105-12. doi: 10.1016/j.nedt.2003.10.001. PMID 14769454
- [Background] Sjostrom-Strand A, Terp K. Parents' Experiences of Having a Baby With a Congenital Heart Defect and the Child's Heart Surgery. Compr Child Adolesc Nurs. 2019 Mar;42(1):10-23. doi: 10.1080/24694193.2017.1342104. Epub 2017 Aug 8. PMID 28786702
- [Background] Johnsson, B.A., M. Nordahl, and B. Magnusson, Evaluating a Dynamic Keep-Alive Messaging Strategy for Mobile Pervasive Systems. Procedia Computer Science, 2017. 109: p. 319-326.
- [Background] Johnsson, B. and B. Magnusson, Supporting Collaborative Healthcare Using PalCom - The itACiH System, in Seventh International Workshop on Pervasive Collaboration and Social Networking. 2016: Sydney, Australia.
- [Background] Holmberg, R., et al., Leadership and implementation of evidence-based practices. . Leadership in Health Services, 2008. 21(3): p. 168-184.
- [Background] Phares V, Lopez E, Fields S, Kamboukos D, Duhig AM. Are fathers involved in pediatric psychology research and treatment? J Pediatr Psychol. 2005 Dec;30(8):631-43. doi: 10.1093/jpepsy/jsi050. Epub 2005 Mar 16. PMID 15772363
- [Background] Heckman JJ. The developmental origins of health. Health Econ. 2012 Jan;21(1):24-9. doi: 10.1002/hec.1802. PMID 22147625
- [Derived] Foldager Jeppesen S, Vilhjalmsson R, Avik Persson H, Kristensson Hallstrom I. Parental satisfaction with paediatric care with and without the support of an eHealth device: a quasi-experimental study in Sweden. BMC Health Serv Res. 2024 Jan 9;24(1):41. doi: 10.1186/s12913-023-10398-7. PMID 38195486
- [Derived] Derwig M, Lindkvist RM, Hallstrom IK, Johnsson BA, Stenstrom P. eHealth usage among parents to premature or surgically treated neonates: associations with eHealth literacy, healthcare satisfaction or satisfaction with an eHealth device. BMC Pediatr. 2023 Oct 21;23(1):524. doi: 10.1186/s12887-023-04340-3. PMID 37865736
- [Derived] Castor C, Lindkvist RM, Hallstrom IK, Holmberg R. Health Care Professionals' Experiences and Views of eHealth in Pediatric Care: Qualitative Interview Study Applying a Theoretical Framework for Implementation. JMIR Pediatr Parent. 2023 Oct 18;6:e47663. doi: 10.2196/47663. PMID 37851500
- [Derived] Hylen M, Nilsson S, Kristensson-Hallstrom I, Kristjansdottir G, Stenstrom P, Vilhjalmsson R. Access to health care perceived by parents caring for their child at home supported by eHealth-a directed approach introducing aperture. BMC Health Serv Res. 2022 Aug 8;22(1):1008. doi: 10.1186/s12913-022-08398-0. PMID 35941653
- See also: World report on disability. — http://www.who.int/disabilities/world_report/2011/en/